CLINICAL TRIAL: NCT02703142
Title: Endoscopic Evaluation for the Postoperative Condition After Esophagectomy and Reconstruction
Brief Title: Endoscopic Evaluation After Esophagectomy
Status: Completed | Type: Observational
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Assistant professor, Nagasaki University
Other Study IDs: NagasakiU
Record Dates: First submitted 2016-01-18; First posted 2016-03-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Neoplasms; Constriction; Anastomotic Leak; Ischemia
Keywords: esophagogastrostomy; gastric conduit ischemia; endoscopy
MeSH Terms: conditions — Esophageal Neoplasms; Constriction, Pathologic; Anastomotic Leak; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dmp-DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients after esophagectomy: Endoscopic examinations are performed at 1, 8, and 15 postoperative days. Endoscopic examination is added when abnormal findings are demonstrated.
  Interventions: Procedure: Patients after esophagectomy

INTERVENTIONS:
Procedure: Patients after esophagectomy — postoperative endoscopic evaluation

SUMMARY:
Gastric conduit ischemia or anastomotic breakdown after esophagectomy with cervical esophagogastrostomy often cause severe complications, such as leakage, necrotic organs, and strictures. Thus, the purpose of this study is the safety and efficacy of endoscopic evaluation about reconstructive organs after esophagectomy. The investigators evaluate endoscopic predictions using classifications in acute phase after esophagogastrostomy.

DETAILED DESCRIPTION:
Gastric conduit ischemia or anastomotic breakdown after esophagectomy with cervical esophagogastrostomy often cause severe complications, such as leakage, necrotic organs, and strictures. However the evaluation and prevention before developing gastric conduit ischemia have been established. The investigators have built a hypothesis that the evaluation for gastric mucosal ischemia in early phase after esophagectomy predict the complication of gastric conduit. Thus, the purpose of this study is the safety and efficacy of endoscopic evaluation about reconstructive organs after esophagectomy. The investigators evaluate endoscopic predictions using classifications in acute phase after esophagogastrostomy.

ELIGIBILITY:
Inclusion Criteria:

* Malignant or end-stage benign esophageal disease.
* Esophagectomy with reconstruction by a gastric pull-up.

Exclusion Criteria:

* Severe heart failure and pulmonary dysfunction
* Severe renal and liver dysfunction
* Allergenic history
* Pregnancy

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo an esophagectomy with reconstruction by a gastric pull-up for malignant or end-stage benign esophageal disease. The patients have a cervical esophagogastrostomy.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with endoscopy-related adverse events as assessed by Clavien-Dindo Classification | From 1 to 29 days after esophagectomy
Number of participants with the classification of gastric conduit ischemia by endoscopic findings | From 1 to 15 days after esophagectomy
Number of participants with the major complications of gastric conduit (strictures, leakage, necrosis) | From 1 to 29 days after esophagectomy

SECONDARY OUTCOMES:
Biological examination of the mucosal biopsy of gastric conduit as assessed by the ischemia related RNA copy number | From 1 to 29 days after esophagectomy
Biological examination of the mucosal biopsy of gastric conduit as assessed by the scoring system for immunohistochemical staining | From 1 to 29 days after esophagectomy
  The scoring system refer to the article entitled a scoring system for immunohistochemical staining: consensus report of the task force for basic research of the EORTC-GCCG. European Organization for Research and Treatment of Cancer-Gynaecological Cancer Cooperative Group (J Clin Pathol. 1997 Oct; 50(10): 801-804.)
Biological examination of gastric conduit as assessed by the Mitochondrial DNA copy number | From 1 to 29 days after esophagectomy

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Kobayashi, Study Director — Department of Surgery, Nagasaki University Graduate School of Biomedical Sciences,
Locations (1):
- Nagasaki University Hospital, Nagasaki, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Protocol information in University Hospital Medical Information Network (UMIN) （UMIN000019585） — https://upload.umin.ac.jp/cgi-open-bin/ctr/ctr.cgi?function=brows&action=brows&type=summary&recptno=R000022640&language=J